CLINICAL TRIAL: NCT05259579
Title: Anti-reflux Mucosal Ablation (ARMA) for the Treatment of Postoperative Gastroesophageal Reflux After Sleeve Gastrectomy - A Pilot Study
Brief Title: ARMA for Postoperative GERD After Sleeve Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Stephen K.K. Ng, Principal Investigator, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2021.553
Record Dates: First submitted 2022-01-26; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anti-reflux mucosal ablation (Experimental): This technique creates an anti-reflux mechanism by performing mucosal ablation at the gastric cardia and inducing cicatrisation, and thereby rebuilds the flap valve at the gastric cardia
  Interventions: Procedure: Anti-reflux mucosal ablation

INTERVENTIONS:
Procedure: Anti-reflux mucosal ablation — Mucosal ablation is planned around the cardia on the gastric side in a butterfly shape. Submucosal layer is raised by injecting saline with indigo carmine dye. Mucosal ablation is performed using the triangle-tip knife in spray coagulation mode.
  Other Names: ARMA

SUMMARY:
This study is a pilot trial designed to evaluate the safety and efficacy of endoscopic anti-reflux ablation in postoperative gastroesophageal reflux after sleeve gastrectomy

ELIGIBILITY:
Inclusion Criteria:

* Patients with reflux symptoms after sleeve gastrectomy and are dependent on or refractory to PPI treatment
* Pathological esophageal acid exposure, defined by DeMeester score >14.7 or acid exposure time (AET) >4.2% on pH study

Exclusion Criteria:

* Primary esophageal motility disorders
* Sliding hiatal hernia >3cm
* Narrow gastric sleeve that precludes retroflexion of scope
* Gastric sleeve stricture
* Malignancy
* Pregnancy
* Patients not fit for general anesthesia
* Other cases deemed by the examining physician as unsuitable for safe treatment
* Refusal to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in GERD symptoms | 3 and 6months
  Gastroesophageal Reflux Disease-Health-Related Quality of Life (GERD-HRQL) questionnaire score [0-75, higher scores mean worse outcome]
Change in GERD symptoms | 3 and 6months
  astroesophageal Reflux Disease Questionnaire (GERDQ) score [0-18, higher scores mean worse outcome]

SECONDARY OUTCOMES:
Technical success rate | 1 day
  defined as successful completion of endoscopic procedure
Change in DeMeester score and AET | 3 months
  evaluated by 24-hour pH monitoring
Dysphagia symptoms | 3 and 6 months
  evaluated by the Brief Esophageal Dysphagia Questionnaire (BEDQ) score [0-40, higher score mean worse outcome]
PPI use | 3 and 6 months
  dosage of PPI use after procedure
Changes in cardia morphology | 3 months
  endoscopic assessment of Hill's flap grade
Adverse events rate relating to endoscopic intervention | 7 days, 1, 3 and 6 months
  complication including bleeding, perforation and stricture

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided